CLINICAL TRIAL: NCT01173081
Title: The Use of Teriparatide as an Adjunctive Therapy for the Treatment of Jones Fractures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ohio Orthopedic Center of Excellence (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B3D-US-X026
Record Dates: First submitted 2010-07-28; First posted 2010-07-30 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Fractures
Keywords: Jones fracture; fifth metatarsal fracture; teriparatide; fracture healing
MeSH Terms: conditions — Fractures, Bone | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teriparatide (Experimental): Patients randomized into this group will inject 20mcg of teriparatide once daily for 16 weeks or until the study endpoint is achieved. Additionally, patients will take oral calcium (1,000mg) and vitamin D3 (1,000 IU) supplements daily.
  Interventions: Drug: Teriparatide
- Placebo Control (Placebo Comparator): Patients randomized into this group will inject a matching dose of placebo once daily for 16 weeks or until the study endpoint is achieved. Additionally, patients will take oral calcium (1,000mg) and vitamin D3 (1,000 IU) supplements daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Teriparatide — 20mcg once daily for 16 weeks or until study endpoint is achieved.
  Other Names: Forteo
  Arms: Teriparatide
Drug: Placebo — matching dose of 20mcg of placebo once daily for 16 weeks or until study endpoint is achieved
  Arms: Placebo Control

SUMMARY:
This randomized, placebo-controlled study will evaluate the effectiveness of the adjunctive use of teriparatide for the healing of Jones fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years of age and who have closed epiphyses.
* Patients of both genders and all races.
* Patients with Jones fractures of the fifth metatarsal less than 2 weeks prior to presenting for clinical evaluation.
* Patients with a history of an acute injury and an acute Jones fracture defined by Torg et al as a fracture line with sharp margins without widening, absence of intramedullary sclerosis, and minimal or no cortical hypertrophy or evidence of periosteal changes due to chronic stress.
* Patients with either no prodromal symptoms or prodromal symptoms present less than 2 weeks.
* Patients with a baseline visual analog scale (VAS) pain score ≤ 20 (100mm scale) for the fifth metatarsal, with the foot at rest and not bearing weight.
* Patients who are in good general health and who have physical examinations that either are within normal limits or are clinically non-significant as determined by the investigator.
* Patients with laboratory evaluations that either are within normal limits or are clinically non-significant as determined by the investigator.
* Patients who have voluntarily signed informed consent forms, including HIPAA Authorization.

Exclusion Criteria:

* Patients who are younger than 18 years of age or patients who are 18 years of age or older with open epiphyses.
* Patients with Jones fractures of the fifth metatarsal greater than 2 weeks prior to presenting for clinical evaluation.
* Patients with tuberosity avulsion fractures or fifth metatarsal shaft fractures.
* Patients with prior fifth metatarsal fracture(s).
* Patients with prodromal symptoms present for more than 2 weeks.
* Patients with a nonunion or delayed union as defined by the radiographic criteria described by Torg et al.
* Patients who are allergic to any of the individual active ingredients in teriparatide or related compounds.
* Patients with chronic rheumatologic disease, ankylosing spondylitis or other inflammatory arthropathy.
* Patients with associated injuries considered by the investigator as to likely interfere with evaluation of the study drug.
* Patients with a present condition or history of any clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematologic, endocrine, neurologic, psychiatric, connective tissue, respiratory or other medical disorders.
* Patients with Worker's Compensation claim(s) under dispute or mediation.
* Patients with history of drug or alcohol abuse.
* Patients who are pregnant or lactating.
* Patients who are considered by the investigator for any reason to be an unsuitable candidate for receipt of the study drug.
* Patients who are unwilling or unable to follow the follow-up evaluation schedules.
* Patients who refuse to voluntarily sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2010-07; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Fracture healing | weeks 4 through 24 after start of treatment

SECONDARY OUTCOMES:
Pain | weeks 4 through 24 after start of treatment
Range of Motion | weeks 4 through 24 after start of treatment
Function | weeks 4 through 24 after start of treatment
Return to Activity | weeks 4 through 24 after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter H. Edwards, Jr., MD, Principal Investigator — Ohio Orthopedic Center of Excellence
Locations (1):
- Ohio Orthopedic Center of Excellence, Upper Arlington, Ohio, United States